CLINICAL TRIAL: NCT03138122
Title: The Study of Men Born in 1943 - A Longitudinal Cohort Study From Middle-Age and Onward
Brief Title: The Study of Men Born in 1943
Status: Active, not recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per-Olof Hansson, M.D, Ph.D.,, Sahlgrenska University Hospital
Other Study IDs: SahlgrenskaUH/Östra
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Risk Factor; Atrial Fibrillation; Congestive Heart Failure; Sleep Apnea; Cardiovascular Diseases
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Sleep Apnea Syndromes; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A random sample a random sample of half of all men born in 1943 and living in the city of Gothenburg, Sweden, have been investigated in 1993 at 50 years of age and will be followed continuously with repeated re-examinations and follow-up concerning mortality and cardiovascular diseased. Out of 1463 invited men, 798 (54.5%) accepted the invitation and is included in this longitudinal cohort study.

DETAILED DESCRIPTION:
In January 1993 a random sample of half of all men born in 1943 and living in the city of Gothenburg, Sweden, was selected and invited to participate a longitudinal observational cohort study. Out of 1463 invited men, 798 (54.5%) accepted the invitation and were examined for 1st time between February 1993 and June 1994. All participants, at 50 years of age, underwent a physical examination including anthropometric measurements, blood pressure and ECG. Several questionaires about previous diseases, life style, physical stress, family history, medications, symptoms and psychosocial factors were included. Blood samples were drawn from an antecubital vein after a nights fast. Basal laboratory analysis were performed. In addition several samples of whole blood, serum and plasma were stored in a freezer (-80○ Celsius) for later analysis.

In 2003, at 60 years of age, a 2nd examination was performed with similar methodology and examination´s. At this time 655 of the original 798 men participated.

A 3rd examination was performed between May 2014 and December 2014. In addition to physical examinations, questionnaires and laboratory analysis an echocardiographic examination, a sleep recording, screening for atrial fibrillation with thumb-EKG and investigation with Arteriography was added.

Echocardiographic examinations were performed by experienced cardiologist in accordance with clinical routine using ultrasound system (Vivid 7 Dimension, GE Medical systems, Horten, Norway), together with commercially available analysis software (GE Vingmed Ultrasound EchoPAC PC, General Electric Healthcare, Little Chalfont, UK) and in agreement with ESC guideline for echocardiography EAE recommendations.

The sleep recording was conducted for one night in the patients home using Apnélink, Apnélink plus or Apnélink air. All participants also answered the Epworth sleepiness scale (ESS) and the functional outcome of sleep questionnaire (FOSQ).

Screening for atrial fibrillation were performed using a thumb-ECG (Zenicor Medical System, Sweden), during a two week-period immediately after the physical examination. ECG was registered by the participants at their home, by placing their thumbs on two electrodes for 30 seconds two times a day, one time in the morning and one in the evening, and also additionally in case they experience any symptoms such as dizziness or palpitations, in a duration of a 2-week period.

In Sweden, all hospital admissions since 1978 are registered in the National Patient Register (NPR) and classified according to the International Classification of Diseases (ICD 8 until 1986; ICD 9 until 1996, ICD 10 since 1997 and continuing). At each examination, information about hospitalizations, medication and morbidity was obtained. During follow-up, death certificates, autopsy reports, and medical records were obtained and studied for all participants. Follow-up will be continues for each of the original 798 participants until death. New examinations will be performed every 5-10 years during follow-up.

Endpoints that are registered include: death, cause of death, myocardial infarction, ischemic heart disease, heart failure with reduced, mid-range and preserved ejection fraction, atrial fibrillation, cerebral infarction, cerebral haemorrhage, diabetes mellitus, deep vein thrombosis, pulmonary embolism, any cancer, fractures and dementia.

The study complies with the Declaration of Helsinki, and the study protocols was approved by the Ethical Committee of Gothenburg (DNR 157-93 in 1993, DNR: 67-03, in 2003 and DNR 649-13 in 2013).

Aims:

1. To study the incidence and prevalence of cardiovascular risk factors and cardiovascular diseases in a random sample from the general population.
2. To study secular trends in cardiovascular risk factors and cardiovascular diseases by comparing this cohort of men born in 1943 to other cohorts of men born in 1913, 1923, 1933, 1953 and 1963 living in the same geographic area and investigated using the same methodology.
3. To study risk factors for various cardiovascular diseases in a longitudinal cohort study.

   In 2016 all men who participated in the 2014 examiniation was invited to a cognitive screening. In total 333 of these men particpated in the screening which included the following tests: Immediate and Delayed Text Recall, Symbol Digit Modalities Test (SDMT), reduced version of The Boston Naming Test, The Clox and Cube Test, The Token Test, Stroop III, Ray-Osterrieth Complex Figure Test (ROCF), F-A-S verbal fluency test. Parallel Serial Mental Operations (PaSMO), and Trailmaking A.

   An additional aim was then added:
4. To study risk factors for dementia / cognitive impairment

ELIGIBILITY:
Inclusion Criteria:

* Men born in 1943 and living in the city of Gothenburg, Sweden

Exclusion Criteria:

* None

Ages: 50 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: A random population sample consisting half of all men born in 1943 and living in the city of Gothenburg, Sweden was invited. . Out of 1463 invited men, 798 (54.5%) accepted participation.
Sampling Method: Probability Sample
Enrollment: 798 (Actual)
Dates: Start 1993-02-09 (Actual); Primary Completion 2043-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular diseases | from date of first examination until the date of endpoint or date of death from any cause, whichever come first assessed up to 20, 30, 40 and 50 years
  Alla major cardiovascular events including cardiovascular death, myocardial Infarction, congestive heart failure atrial fibrillation, stroke and venous thromboembolism

SECONDARY OUTCOMES:
Sleep apnoea syndrome | at 71 years of age
  Apnoea and hypopnoea as well as desaturation defined according to guide lines for scoring sleep apnoea.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital / Östra, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barywani SB, Ostgard Thunstrom E, Mandalenakis Z, Hansson PO. Body iron stores had no impact on coronary heart disease outcomes: a middle-aged male cohort from the general population with 21-year follow-up. Open Heart. 2022 Apr;9(1):e001928. doi: 10.1136/openhrt-2021-001928. PMID 35410912
- [Derived] Sakalaki M, Hansson PO, Rosengren A, Thunstrom E, Pivodic A, Fu M. Multi-modality biomarkers in the early prediction of ischaemic heart disease in middle-aged men during a 21-year follow-up. BMC Cardiovasc Disord. 2021 Feb 2;21(1):65. doi: 10.1186/s12872-021-01886-x. PMID 33530933
- [Derived] Chen X, Thunstrom E, Hansson PO, Rosengren A, Mandalenakis Z, Zhong Y, Ergatoudes C, Caidahl K, Fu M. High prevalence of cardiac dysfunction or overt heart failure in 71-year-old men: A 21-year follow-up of "The Study of men born in 1943". Eur J Prev Cardiol. 2020 May;27(7):717-725. doi: 10.1177/2047487319871644. Epub 2019 Aug 25. PMID 31446787